CLINICAL TRIAL: NCT00641953
Title: A Randomized, Phase II, Multi-Center, Double-Blind, Placebo-Controlled, Dose-Response Study of an Aqueous Topical Formulation of Nitroglycerin, IMX-150, in the Treatment of Pain in Diabetic Peripheral Neuropathy of the Feet
Brief Title: IMX-150 Cream for Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Procris Pharmaceuticals (Industry)
Responsible Party: Matthew A. Gonda, PhD, Procris Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-004A
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Foot Pain; Diabetic Neuropathy Pain; Diabetic Peripheral Neuropathy foot pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): IMX-150 (0.3%) 0.5 g topically BID each foot
  Interventions: Drug: IMX-150
- B (Experimental): IMX-150(0.6%) 0.5 g topically BID to each foot
  Interventions: Drug: IMX-150
- C (Placebo Comparator): Placebo 0.5 g topically BID to each foot for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IMX-150 — (0.3%) 0.5g topically BID to each foot for 4 weeks
  Arms: A
Drug: IMX-150 — (0.6%) 0.5g topically BID to each foot for 4 weeks
  Arms: B
Drug: Placebo — 0.5 g topically BID to each foot for 4 weeks
  Arms: C

SUMMARY:
The purpose of this study is to compare the effectiveness of two different dose of IMX-150 to that of placebo (non-active) in the treatment of diabetic peripheral neuropathy pain of the feet.

ELIGIBILITY:
Inclusion Criteria:

* Must have sufficient command and understanding of the English language to complete diaries and questionnaires
* If female, may not be pregnant or lactating
* Can be treated on an outpatient basis
* Has a clinical diagnosis of Type-1 or Type II diabetes with: confirmed diagnosis of diabetic distal symmetrical sensorimotor polyneuropathy and bilateral pain in the feet for at least 3 months.
* Must have a hemoglobin A1C value of 11% or less that is stable under treatment
* Agrees to use the test creams as specified for the 4 week period
* Willing to not use any other medications, including investigational medications, to treat pain symptoms of Diabetic Neuropathy while in study.

Exclusion Criteria:

* Currently using any nitrate medications
* Currently using Viagra®, Levitra®, Cialis® or other phosphodiesterase 5 inhibitors medications for erectile dysfunction
* Currently treated for symptoms of diabetic neuropathy, including but not limited to Lyrica®, Cymbalta® and transcutaneous stimulation
* Not on a stable dose for at least 4 weeks prior to study screening of other vasodilators required for underlying conditions
* Know allergy to Nitroglycerin, propylene glycol or common moisturizing creams
* History of migraine, cluster or vascular headaches, chronic pain with greater pain intensity than the pain of diabetic neuropathy or other chronic pain condition within the region of the diabetic peripheral neuropathy
* Amputation of more than one toe per foot
* Neurological disorder or skin condition that may alter local sensation in the feet
* History of unstable medical problem, clinically significant screening laboratory test or any current medical condition that would contraindicate the administration of the study mediation, interfere with the study evaluations, or interfere with the patient's ability to comply with the study
* History of drug (including cannabinoid) or alcohol abuse within the past year
* Cognitive or language difficulties that would impair completion of the pain assessment tool
* Within the past 3 months, have had either a myocardial infarction, uncontrolled hypotension, or uncontrolled hypertension
* Participated in a study of any investigational drug within 4 weeks or 5 half-lives of the drug, whichever is longer, prior to Screening
* Major abdominal, thoracic or vascular surgery within 6 months of the first dose of study medication
* Open lesions in the area where the cream is to be applied
* Fertile patients who are unable or unwilling to comply with the contraceptive requirements during the study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2007-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to endpoint (Day 29) in the average of neuropathic foot daily pain "24 - Hour Average Pain" scores | Weekly average of "24-hour Average Pain"

SECONDARY OUTCOMES:
Change in weekly average sleep disturbance | daily

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Yeramian, MD, Study Director — VP Medical Affairs
Locations (7):
- United States (7):
  - Meriden Research, Brooksville, Florida
  - Health Awareness, Jupiter, Florida
  - International Research Associates, LLC, Miami, Florida
  - Peninsula Research, Ormond Beach, Florida
  - Alpha Medical Research, Oviedo, Florida
  - Meridien Research, St. Petersburg, Florida
  - Hampton Roads Center for Clinical Research, Norfolk, Virginia